CLINICAL TRIAL: NCT06842745
Title: Personalized Transcranial Magnetic Stimulation and Constraint Induced Language Therapy to Treat Mild Post-Stroke Aphasia
Brief Title: Transcranial Magnetic Stimulation + Language Therapy to Treat Mild Aphasia
Acronym: TMS
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: University of Pennsylvania (Other)
Collaborators: Temple University (Other); National Institute on Deafness and Other Communication Disorders (NIDCD) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 857363; 1R21DC021833-01 (NIH)
Record Dates: First submitted 2025-02-18; First posted 2025-02-24 (Actual); Last update posted 2025-02-24 (Actual); Status verified 2025-02

CONDITIONS: Aphasia; Stroke; Aphasia Following Cerebral Infarction; Aphasia, Acquired
Keywords: aphasia; stroke; non-invasive brain stimulation; Transcranial Magnetic Stimulation
MeSH Terms: conditions — Aphasia; Stroke | interventions — Transcranial Magnetic Stimulation; Speech Therapy

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Real TMS (Experimental): Some of our participants will be randomized to the real treatment arm where they will receive 10 sessions of real TMS paired with speech-language therapy.
  Interventions: Device: Transcranial Magnetic Stimulation (TMS); Behavioral: Speech-Language Therapy (SLT)
- Fake TMS (Sham Comparator): Some of our participants will be randomized to the sham treatment arm where they will receive 10 sessions of fake TMS paired with speech-language therapy.
  Interventions: Behavioral: Speech-Language Therapy (SLT)

INTERVENTIONS:
Device: Transcranial Magnetic Stimulation (TMS) — TMS, is a form of non-invasive brain stimulation, that uses magnetic pulses to stimulate specific areas of the brain. In this study we will utilize theta-burst stimulation which uses a higher frequency pulse of 50 Hz delivered for 40 seconds for a total of 600 pulses.
  Arms: Real TMS
Behavioral: Speech-Language Therapy (SLT) — Our SLT protocol draws from two theories and evidence-based cognitive-linguistic frameworks: (1) conversational alignment, which engages priming of lexical and syntactic structures through dialogue and conversation and (2) increased tolerance of memory load in the context of sentence repetition and dialogue tasks. Administration of these tasks will abide by principles of constraint-induced language therapy, i.e., intense treatment schedule and verbal responding only.
  All participants will receive SLT.

SUMMARY:
The goal of this clinical trial is to determine if Transcranial Magnetic Stimulation (TMS) combined with Speech-Language Therapy (SLT) is an effective treatment for mild aphasia in persons with chronic stroke.

The main questions this study aims to answer are:

1. Can TMS combined with SLT improve conversational speech and comprehension?
2. Can we identify specific behavioral and biological characteristics that would benefit most from the TMS and SLT treatment?

Researchers will compare real TMS to sham (fake) TMS to see whether TMS can treat post-stroke mild aphasia.

Participants will:

* Complete a screening and medical intake to determine eligibility
* Undergo a MRI
* Participate in 10 consecutive sessions (Monday-Friday) of TMS and SLT treatment
* Complete follow-up assessments 2 and 4 months after treatment

DETAILED DESCRIPTION:
Aphasia is an acquired disorder of language that occurs in approximately 30% of individuals with stroke and impacts approximately 1 million Americans (see NINDS.NIH.gov). Current treatments for aphasia are only modestly beneficial, so there is a clear need for more efficacious therapy.

Previous research has demonstrated that TMS improves language performance in persons with aphasia and the benefit has been shown to be sustained. All studies of which we are aware, however, have included participants with moderate/severe aphasia. The issue of mild aphasia has received little attention to date but as there is an increasing recognition that even very mild language deficits have important negative consequences for employment and social well-being. This study will aim to treat mild aphasia with TMS and SLT emphasizing conversations speech.

One limitation of TMS has been variability in response; TMS has shown good within-subject reliability but more substantial variability between subjects. In recognition of these issues, "electrical field" (e-field) models have been developed to account for these individual differences in anatomy. We will the utilize e-field models in conjunction with an individually determined resting motor threshold to generate a personalized treatment regimen that is likely to ensure that all subjects receive the same TMS intensity relative to their individual motor threshold and greatly reduces the possibility of under- or over-dosing with respect to TMS intensity. We will employ continuous theta-burst stimulation, 600 brief electrical pulses delivered in 40 seconds, over the right front part of the brain (pars triangularis).

Participants who are enrolled can expect to undergo a battery of tests to define their language function as well as a research MRI scan that will be used to guide TMS therapy and to assess the size and location of the stroke and its impact on brain pathways. After baseline testing, subjects will undergo treatment using TMS (or sham) + SLT for 10 sessions (Monday-Friday) over the course of 2 consecutives week. Follow-up assessment of language functioning will be assessed immediately, 2 months and 4 months after treatment.

Participants will be compensated for their time and travel.

ELIGIBILITY:
Inclusion Criteria:

* Left Hemisphere stroke
* Stroke occurred more than 6 months ago
* Mild Aphasia (WAB AQ score > 85)
* Proficient in English

Exclusion Criteria:

* Ongoing substance or alcohol abuse
* Other neurological disorders, beside stroke (i.e. dementia, traumatic brain injury, multiple sclerosis)
* Active psychiatric disorders (i.e. bipolar disorder, schizophrenia)
* Pacemaker or cardiac defibrillator
* Diagnosis of tinnitus
* Epilepsy, or seizure in the past 6 months

Ages: 40 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 24 (Estimated)
Dates: Start 2025-02-11 (Actual); Primary Completion 2026-08-31 (Estimated); Study Completion 2026-08-31 (Estimated)

PRIMARY OUTCOMES:
Sentence Processing | From baseline to 4 months post-intervention
  Change in performance on the Temple Assessment of Language and Short-term Memory in Aphasia (TALSA) sentence processing composite score.

SECONDARY OUTCOMES:
Semantic and Phonological Processing | From baseline to 4 months post-intervention
  Change in performance on the TALSA composite semantic processing score and phonological processing score.
Elicited Speech | From baseline to 4 months post-intervention
  Change in performance on the Nicholas & Brookshire picture description and Story Retell scores.

CONTACTS AND LOCATIONS:
Overall Officials: H. Branch Coslett, MD, Principal Investigator — University of Pennsylvania
Locations (1):
- University of Pennsylvania, Philadelphia, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: No
No, the study team does not plan to share participating data at this time.